CLINICAL TRIAL: NCT06315205
Title: A Phase I, Open Label, Dose Escalation Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Single Intramuscular Injections of Letrozole LEBE at Different Strengths in Voluntary Healthy Post-Menopausal Women.
Brief Title: Evaluation of the Pharmacokinetics, Safety, and Tolerability of IM Letrozole LEBE in Healthy Post-menopausal Women
Acronym: LEILA-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ROV-LEBE-2023-01; 2023-503948-13 (EudraCT Number)
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Safety; Letrozol LEBE; Intramuscular; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Letrozol LEBE 75 mg (Experimental)
  Interventions: Drug: Letrozole LEBE 75 mg
- Cohort 2: Letrozol LEBE 150 mg (Experimental)
  Interventions: Drug: Letrozole LEBE 150 mg
- Cohort 3: Letrozol LEBE 225 mg (Experimental)
  Interventions: Drug: Letrozole LEBE 225 mg

INTERVENTIONS:
Drug: Letrozole LEBE 75 mg — 14 oral doses of Femara 2.5 mg/daily + 28-days (at least) washout period + single IM injection of Letrozole LEBE 75 mg
  Arms: Cohort 1: Letrozol LEBE 75 mg
Drug: Letrozole LEBE 150 mg — 14 oral doses of Femara 2.5 mg/daily + 28-days (at least) washout period + single IM injection of Letrozole LEBE 150 mg
  Arms: Cohort 2: Letrozol LEBE 150 mg
Drug: Letrozole LEBE 225 mg — 14 oral doses of Femara 2.5 mg/daily + 28-days (at least) washout period + single IM injection of Letrozole LEBE 225mg
  Arms: Cohort 3: Letrozol LEBE 225 mg

SUMMARY:
This is a Phase I, open label, sequential, single ascending dose (SAD) study to evaluate the pharmacokinetic (PK), safety, and tolerability of Letrozole LEBE in healthy post-menopausal women.

DETAILED DESCRIPTION:
The study consists of 1 Screening Period and 2 treatment periods. Evaluation of eligibility and allocation of subject number to the volunteers will be performed after Screening. It is planned that subjects will be enrolled in three groups of approximately 30 subjects in each group (Groups 1 to 3), in order to ensure 15 completed subjects per group in Treatment Period 1 and Treatment Period 2. In Treatment Period 1, each subject will sequentially receive 1 dose daily of oral Femara (2.5 mg) over a period of 14 days followed by a single intramuscular (IM) dose of Letrozole LEBE (after a washout period) in Treatment Period 2. Ascending doses of Letrozole LEBE will be given to Groups 1, 2 and 3. Safety and tolerability will be assessed in all groups by the incidence and severity of Adverse Events (AEs) and Serious AEs (SAEs), concomitant medication use, vital sign assessments, clinical laboratory evaluations, 12 lead ECGs, physical examination, and body weight/BMI. The end of the clinical trial will be the last visit of the last subject at Day 197 of Treatment Period 2 or any additionally required 4-weeks safety follow up visits, when plasma levels of letrozole are detectable, whichever occurs later. Those remaining subjects with detectable plasma levels of letrozole could be followed every 4 weeks.

The sample size was estimated based on a minimum number necessary to obtain a preliminary assessment regarding the drug's PK and safety profile over the planned dose range. No formal sample size calculation was made for this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy post-menopausal women.
* Capable of providing informed consent.
* Weight of ≥50 kg and a BMI ≥19 and ≤39 kg/m2.
* Subjects should be able to communicate with clinic staff.

Exclusion Criteria:

* Subjects who have a history of allergy or hypersensitivity to letrozole or any of the inactive ingredients.
* Subjects who have a history of galactose intolerance, severe hereditary lactase deficiency glucose-galactose malabsorption.
* Subjects who have used estrogen or progesterone hormone replacement therapy, thyroid replacement therapy, oral contraceptives, androgens, luteinizing hormone (LH) releasing hormone analogs, prolactin inhibitors, or antiandrogens within prior to Screening.
* Subjects who have used: any medications including St. John's wort or any medications or products known to be potent or moderate inhibitors of CYP P450 3A4.
* Subjects who have been diagnosed with osteoporosis.
* Subjects who have an abnormality at Screening or prior to first dose that in the opinion of the investigator increases the risk of participating in the study.
* Subjects who have any clinically significant abnormal physical examination or laboratory safety findings at screening.
* Subjects who have relevant diseases or clinically significant abnormal relevant findings at Screening, as determined by medical history, physical examination, laboratory, ECG, DEXA, and breast and pelvic examination.
* Subjects who have history of any significant chronic disease.
* History of cancer within the past 5 years with the exception of non-melanoma skin cancer.
* Subjects who have a history of drug-dependence, and recent history of alcoholism or abuse of alcohol.
* Subjects who have received a drug in research or have participated in other clinical trials within 90 days, prior to dosing.
* Any other unspecified reason that, in the opinion of the investigator (or designee) or sponsor, makes the subject unsuitable for enrolment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
λz | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Terminal phase elimination rate constant
Cmax | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Maximum observed plasma concentration after Letrozole LEBE administration
Clast | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Last observed plasma concentration after Letrozole LEBE administration
tmax | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Time to maximum observed concentration
tlag | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Lag time before observation of quantifiable concentrations in plasma.
t1/2 | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Terminal elimination half life.
AUC∞ | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Area under the concentration time curve from time zero extrapolated to infinity.
AUClast | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Area under the concentration time curve from time zero up to the last quantifiable concentration.

SECONDARY OUTCOMES:
E1 | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Estrone
SE1 | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Sulfate estrone
E2 | Following single IM administration of Letrozole LEBE (Treatment Period 2, Day 1) until Day 197
  Estradiol
λz | Following multiple oral administration of Femara (Treatment Period 1, Day 14)
  Terminal phase elimination rate constant.
Cav | Following multiple oral administration of Femara (Treatment Period 1, Day 14)
  Average plasma concentration over a dosing interval.
Cmin, ss | Following multiple oral administration of Femara (Treatment Period 1, Day 14)
  Minimum observed plasma concentration at steady-state.
Cmax,ss | Following multiple oral administration of Femara (Treatment Period 1, Day 14)
  Maximum observed plasma concentration at steady-state
tmax | Following multiple oral administration of Femara (Treatment Period 1, Day 14)
  Time to maximum observed concentration.
t1/2 | Following multiple oral administration of Femara (Treatment Period 1, Day 14)
  Terminal elimination half-life.
AUCτ | Following multiple oral administration of Femara (Treatment Period 1, Day 14)
  Area under the concentration-time curve over a dosing interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site number CZ-01, Prague, Czechia